CLINICAL TRIAL: NCT02796508
Title: Age-related Cognitive Decline: Effects of Video Game Training on Behavioral and Neuroimaging Measures of Attention and Memory
Brief Title: Attention and Memory Training With Video Games in Old Age
Acronym: AGEGAME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional de Educación a Distancia (Other)
Responsible Party: Principal Investigator, Soledad Ballesteros, Professor, Universidad Nacional de Educación a Distancia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PSI2013-41409R
Record Dates: First submitted 2016-05-12; First posted 2016-06-10 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Ageing
Keywords: Healthy aging; Cognitive training; Video-games; Attention; Working memory; Wellbeing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Non-action video game training (Experimental): Experimental: Non-action video game training 16 1-hour training sessions with 10 non-action video game training selected games from Lumosity.
  Interventions: Behavioral: Experimental: Non-action video game training
- Non-cognitive video game training (Active Comparator): Active Control: Non-cognitive social video game training 16 1-hour training sessions with non-cognitive video game training with social games from The Sims.
  Interventions: Behavioral: Active Comparator: Non-cognitive video game training

INTERVENTIONS:
Behavioral: Experimental: Non-action video game training — PSI2013-41409R. Effects of video game training on behavioral and neuroimaging measures of attention and memory
  Other Names: 16 training session with Lumosity over 8-10 weeks in small groups
  Arms: Non-action video game training
Behavioral: Active Comparator: Non-cognitive video game training — 16 training sessions with The Sims over 8-10 weeks in small groups
  Other Names: Social video game training
  Arms: Non-cognitive video game training

SUMMARY:
Neuroplasticity-based approaches seem very promising to maintain cognitive health in older adults and postpone the onset of cognitive-decline and dementia symptoms. The aims of this project are threefold:

1. the evaluation of the effects of a neuroplasticity-based-cognitive randomized computer-based intervention consisting in training with non-action video games on brain and cognitive functions that decline with ageing, including attention and spatial working memory (WM), in older adults using behavioral measures and electrophysiological recordings (event-related potentials -ERPs- and event-related spectral perturbations -ERSPs);
2. the study of the effects of age and 3 months maintenance on the cognitive and neural signatures of transfer effects to attentional and spatial WM tasks; and
3. to investigate the neuroinflammatory mechanisms assessed by non-invasive methods in saliva from participants underlying cognitive training-induced effects.

A better understanding of these mechanisms elucidates pathways that may be targeted in the future, either by behavioral or neuropsychological interventions. To achieve these aims, the investigators will recruit between 60-80 older adults volunteers to participate in the randomized, controlled, single-blind study. After screening, participants will be randomly distributed in one of these two groups: experimental and active control. Participants in the experimental group will receive 16 1 hour computerized training with non-action video games. The active control group will receive 16 1 hour training sessions with a social video game. The design is a mixed factorial design with type of intervention (experimental, active control) and assessment session (pre, post, maintenance). The results from the proposed research project will clarify the existence of transfer-of-benefit and neural mechanisms underlying cognitive improvement. The hypothesis is that mental stimulation through non-action video games will improve attention and memory, promoting brain and mental health, and extending independence among elderly people by avoiding the negative personal and economic consequences of long-term care.

ELIGIBILITY:
Inclusion Criteria:

* Mini-Mental State Examination (MMSE) score 26 or greater
* Global Deterioration Scale (GDS) score less than 5
* Independent living
* Normal or correct to normal vision and hearing

Exclusion Criteria:

* Diagnosis of dementia
* Planned move from study area
* Inability to complete study activities
* Scores lower than inclusion criteria requirements
* Communication problems.

Ages: 55 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
STROOP-Negative Priming | Change from Baseline Stroop-Negative Priming task at 15 weeks and 30 weeks
  Participants with non-action video-game training, change from baseline in selective attention and capacity to inhibit information on Stroop-Negative Priming task at 15 weeks and maintenance at 30 weeks
ODDBALL | Change from Baseline oddball task at 15 weeks and 30 weeks
  Participants with non-action video-game training, change from baseline in alertness and distraction on Oddball task at 15 weeks and maintenance at 30 weeks
N-BACK | Change from Baseline N-back task at 15 weeks and 30 weeks
  Participants with non-action video-game training, change from baseline in working memory on N-back task at 15 weeks and maintenance at 30 weeks
CORSI BLOCK | Participants with non-action video-game training, change from baseline Corsi block task at 15 weeks and 30 weeks
  Participants with video-game training, change from baseline in spatial working memory on Corsi block task after at 15 weeks and maintenance at 30 weeks

SECONDARY OUTCOMES:
Improvement of the performance (accuracy scores) obtained on the non-action video games (experimental group) and the non-cognitive video games (active comparator) comparing accuracy scores of the first to the last training session. | Change from the first training session to the last (16th) training session, up to 12 weeks
  Efficacy of training: Better performance in the trained video games from first to the last training session comparing accuracy scores of the first to the last training session.
Level of motivation assessed with a questionnaire | Maintenance during the 16 training sessions of non-action cognitive video game training and non-cognitive training at first session, 8th and 16th training sessions. Up to 12 weeks.
  Maintenance of motivation from the first to the last training sessions

CONTACTS AND LOCATIONS:
Overall Officials: Soledad Ballesteros, Ph.D., Principal Investigator — Departament of Basic Psychology II, Universidad Nacional de Educación a Distancia (UNED)
Locations (1):
- Department of Basic Psychology II (UNED), Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Ballesteros S, Mayas J, Ruiz-Marquez E, Prieto A, Toril P, Ponce de Leon L, de Ceballos ML, Reales Aviles JM. Effects of Video Game Training on Behavioral and Electrophysiological Measures of Attention and Memory: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2017 Jan 24;6(1):e8. doi: 10.2196/resprot.6570. PMID 28119279
- [Derived] Ballesteros S, Mayas J, Prieto A, Ruiz-Marquez E, Toril P, Reales JM. Effects of Video Game Training on Measures of Selective Attention and Working Memory in Older Adults: Results from a Randomized Controlled Trial. Front Aging Neurosci. 2017 Nov 1;9:354. doi: 10.3389/fnagi.2017.00354. eCollection 2017. PMID 29163136